CLINICAL TRIAL: NCT01958983
Title: The Effect of Music Therapy on Emotion and Cognition for Individuals With Mild to Moderate Dementia
Brief Title: Music Therapy to Promote Emotion and Cognition for Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101-3041B
Record Dates: First submitted 2013-10-06; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-09

CONDITIONS: Dementia
Keywords: dementia; drumming; emotion; cognition; functional MRI
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music Therapy Group Session (Experimental): Participants will receive 60-minute group session twice a week over 2 months of period. Each session will be led by a music therapist. The contents of the music therapy session include drumming, rhythm imitation, score reading, lyrics comprehension, singing, and song discussion.
  Interventions: Behavioral: Music Therapy Group Session
- No Music Therapy Session (No Intervention): Participants will receive pre- and post-assessments and evaluations at 0 and 2 months. No intervention will be provided. Music therapy sessions will be offered to participants in completion of their study participation.

INTERVENTIONS:
Behavioral: Music Therapy Group Session
  Arms: Music Therapy Group Session

SUMMARY:
The purpose of this study is to determine if the effects of music therapy alter emotion and cognition performances of individuals with mild to moderate dementia. The music therapy intervention protocol is structured by drum improvisation, rhythm imitation, music cognition and song discussion. Attentive listening and active participation of the music training activities allow participants to utilize their focus of attention and comprehension of informational texts. Music therapy intervention is proposed to provide positive stimulations on emotion and cognitive functions of individuals with dementia. The results of the present study will clarify relationship between the effect of music therapy and the neural substrate of music therapy in anatomical and functional brain data obtained from MRI (fMRI).

DETAILED DESCRIPTION:
Individuals with dementia often exhibit deterioration in cognitive functions and experience changes in emotions and personalities. Due to the changes in the frontal and temporal lobes of the brain, individuals with dementia often experience an impaired ability to judge situations. Empirical studies have indicated that cognitive stimulation is essential to facilitate individuals with dementia in thinking, concentration, and memory. Structured music activities provide cognitive stimulation to individuals with dementia through attentive listening and active participation. Additionally, drum improvisation not only reflects the current status of an individual, but also serves as an audio feedback through free play.

ELIGIBILITY:
Inclusion Criteria:

* a mild dementia diagnosis with Clinical Dementia Rating (CDR) score: 1 and The Mini Mental State Examination (MMSE) score: 18-24

Exclusion Criteria:

* significant visual and hearing impairment that hinders music listening and score reading
* for fMRI safty: with shrapnel or other metal or electronic implants in their bodies

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Brain Changes from Baseline on Functional and Structural Connectivity at 2 Months by Multi-Model MRI Analyses | Baseline and after 8-week music therapy intervention
  All participants will received two MRI scans at 0 and 2 months. Images will be acquired on a 3.0T Siemens MRI scanner with 12-channels head coil. All the images are acquired parallel to the anterior commissure-posterior commissure line. To minimize motion artifact generated during the image acquisition, each participant's head will be immobilized with cushions inside the coil. Three kinds of MRI techniques will be performed in this study, including T1-weighted high-resolution anatomical image, resting-state function MRI, and half-sphere diffusion spectrum imaging. Therefore, T1VBM(voxel-based morphology), TBSS(tract-based spatial statistics), functional brain network analysis, and structural brain network analysis will be employed for evaluating the changes of brain functional and structural connectivity in individuals with dementia in experimental and control groups.

SECONDARY OUTCOMES:
Change from Baseline on Geriatric Depression Scale (GDS) at 2 Months | Baseline and at 2 Months
Change from Baseline on Cohen-Mansfield Agitation Inventory (CMAI) at 2 Months | Baseline and at 2 Months
Change from Baseline on Inventory of Quality of Life (SF-36) at 2 Months | Baseline and at 2 Months
Change from Baseline on Frontal Assessment Battery (FAB) at 2 Months | Baseline and at 2 Months
Change from Baseline on Quality of Drum Improvisation at 2 Months | Baseline and at 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Pei, PhD, Principal Investigator — Chang Gung Medical Foundation
Locations (1):
- Chang Gung Medical Foundation, Taoyuan District, Taiwan, Taiwan

REFERENCES:
- [Derived] van der Steen JT, van der Wouden JC, Methley AM, Smaling HJA, Vink AC, Bruinsma MS. Music-based therapeutic interventions for people with dementia. Cochrane Database Syst Rev. 2025 Mar 7;3(3):CD003477. doi: 10.1002/14651858.CD003477.pub5. PMID 40049590